CLINICAL TRIAL: NCT05921500
Title: Clinical and Radiographic Evaluation of Intra Coronal Bleaching of Primary Anterior Teeth Using Sodium Perborate With Walking Bleach Technique
Brief Title: Clinical and Radiographic Evaluation of Intra Coronal Bleaching of Primary Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Yasser Mohammed Bedir, cairo, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: internal bleaching
Record Dates: First submitted 2023-06-03; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Dental Trauma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internal bleaching of discolored primary anterior teeth by using sodium peborate (Experimental): Internal bleaching of discolored primary anterior teeth by using sodium peborate
  Interventions: Drug: sodium peborate

INTERVENTIONS:
Drug: sodium peborate — Internal bleaching of discolored primary anterior teeth by using sodium peborate

SUMMARY:
clinical and radiographic evaluation the intracoronal bleaching of primary anterior teeth using sodium perborate with walking bleach technique

DETAILED DESCRIPTION:
This study will be conducted for the clinical and radiographic evaluation the intracoronal bleaching of primary anterior teeth using sodium perborate with walking bleach technique

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3-5 years.
* Parents/caregivers acceptance.
* Traumatized anterior teeth with sensitivity to percussion and palpation with gray discoloration.
* Discolored anterior teeth indicated for intracoronal bleaching.
* Traumatized anterior teeth no response to an electric pulp test.
* Discolored teeth with satisfactorily previously obturated root canal .
* Absence of preapical lesions or apex resorption.

Exclusion Criteria:

* Teeth with signs tooth mobility indicated for extraction.
* Teeth with vertical root fracture.
* Teeth with preapical lesions or apex resorption.
* Teeth with discolorations from restorative materials.
* Children with lack of cooperation for post-operative recall and follow up.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation of internal bleaching of primary teeth | two weeks to month
  Clinical outcomes:
  During the follow-up period- two weeks to month, signs of any pathology will be observed clinically and scored as follow:
  1. Sensitivity to percussion or palpation (positive or negative).
  2. Abscess or fistulae (positive or negative).
  3. Color change recorded by vita shade 3d master.

SECONDARY OUTCOMES:
radiographic evaluation of internal bleaching of primary teeth | six months
  Radiographically outcomes:
  During the follow-up period - six months, signs of any pathology will be observed radiographically and scored as follow:
  1. External or internal root resorption (positive or negative).
  2. Apical radiolucency (positive or negative).

CONTACTS AND LOCATIONS:
Overall Officials: alaa eldin mohamed, associate professor, Study Director — associate professor; hamdy badreldin, lecture, Study Director — lecture
Locations (1):
- Yasser Mohammed Bedir, Tanta, Egypt

REFERENCES:
- [Background] Arikan V, Sari S, Sonmez H. Bleaching a devital primary tooth using sodium perborate with walking bleach technique: a case report. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 May;107(5):e80-4. doi: 10.1016/j.tripleo.2009.01.050. PMID 19426913
- [Background] Sharma DS, Barjatya K, Agrawal A. Intra-coronal bleaching in young permanent and primary tooth with biologic perspectives. J Clin Pediatr Dent. 2011 Summer;35(4):349-52. doi: 10.17796/jcpd.35.4.p372w1h5j2kg5734. PMID 22046690